CLINICAL TRIAL: NCT00389740
Title: A Randomized, Double-Blind, Double-Dummy, Parallel-Group, Multicenter Study to Evaluate and Compare the Effects of Alendronate and Raloxifene on Bone Mineral Density in Postmenopausal Women With Osteoporosis
Brief Title: A Comparison Study With Alendronate and Raloxifene in Postmenopausal Women With Osteoporosis (0217-189)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0217-189; 2006_537
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Last update posted 2024-08-14 (Actual); Status verified 2022-02

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Duration of Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0217, /Duration of Treatment : 12 Months
Drug: Comparator : raloxifene hydrochloride /Duration of Treatment : 12 Months

SUMMARY:
The purpose of this study is to compare how well alendronate and raloxifene increase the bone density in women who have osteoporosis and have experienced menopause.

ELIGIBILITY:
Inclusion Criteria:

* Patient is postmenopausal (or surgically menopausal) for at least 6 months
* Patient must be diagnosed with osteoporosis
* Patient has spinal anatomy suitable for DEXA of the lumbar spine

Exclusion Criteria:

* Patient is receiving or has received treatment prior to randomization which might influence bone turnover
* Patient has a history of or evidence for metabolic bone disease (other than postmenopausal bone loss)
* Patient is receiving or is expected to receive during the course of the study any medication (other than study medication) which might alter bone or calcium metabolism

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2001-04-02 (Actual); Primary Completion 2003-01-16 (Actual); Study Completion 2003-01-16 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density (BMD) in PA lumbar spine at 12 months

SECONDARY OUTCOMES:
Bone Mineral Density (BMD) in hip at 12 months; bone turnover at 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Luckey M, Kagan R, Greenspan S, Bone H, Kiel RD, Simon J, Sackarowitz J, Palmisano J, Chen E, Petruschke RA, de Papp AE. Once-weekly alendronate 70 mg and raloxifene 60 mg daily in the treatment of postmenopausal osteoporosis. Menopause. 2004 Jul-Aug;11(4):405-15. doi: 10.1097/01.gme.0000119981.77837.1f. PMID 15243278